CLINICAL TRIAL: NCT03238638
Title: A Phase II Study of Epacadostat + Pembrolizumab in Head and Neck Cancer Patients, Who Failed Prior PD-1/PD-L1 Therapy
Brief Title: A Study of Epacadostat + Pembrolizumab in Head and Neck Cancer Patients, Who Failed Prior PD-1/PD-L1 Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI did not attempt to open the study.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1631
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Head and Neck Cancer
Keywords: Epacadostat; Pembrolizumab; PD-1; PD-L1
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acquired Resistance Cohort and Suboptimal Benefit Cohort (Experimental): Patients will be divided into two cohorts. Investigators anticipate 15 patients per cohort.
  Cohort 1: Acquired Resistance Cohort
  * Treat upon emergence of acquire resistance
  * Prior benefit from an9-PD-1/PD-L1 therapy defined as a. preior response, and/or b. greater than or equal to 5 months of stable disease
  * Progressive disease on recent scans
  * Intercurrent therapy is allowed
  Cohort 2: Suboptimal Benefit Cohort
  * Treat subop. mal response/benefit, BEFORE emergence of acquired resistance
  * Prolonged stable disease greater than or equal to 5 months OR Subop9mal response (greater than 10% and less than 50%)
  * Ongoing stable disease on recent scans
  Both cohorts will receive pembrolizumab and epacadostat.
  Interventions: Drug: Pembrolizumab; Drug: epacadostat

INTERVENTIONS:
Drug: Pembrolizumab — Both cohorts will receive pembrolizumab at a flat dose of 200mg every 3 weeks.
  Other Names: Keytruda
Drug: epacadostat — Both cohorts will receive epacadostat. Patients in cohort 1 will take 300mg of epacadostat by mouth twice per day. Cohort 2 will take 300mg of epacadostat every 6 weeks.

SUMMARY:
This is a research study to test the combination of two drugs, pembrolizumab and epacadostat with the goal of benefiting subjects with head and neck cancers where prior or ongoing regimens with a PD-1 or PD-L1 inhibitor for the treatment of advanced head and neck cancer after platinum failure.

DETAILED DESCRIPTION:
Primary Objective(s) & Hypothesis

(1) Objective: Response Rate

Hypotheses:

Cohort 1: In patient with prior response to anti-PD-1/PD-L1+ therapy and subsequent (acquired) resistance combined IDO1 and PD-1 inhibition will re-induce responses.

Cohort 2: In patients with suboptimal benefit from prior anti-PD-1/PD-L1 therapy combined IDO1 and PD-1 inhibition will induce clinically meaningful responses.

Secondary Objective(s) & Hypothesis

1. Objective: 1-year Progression-free (PFS) and Overall (OS) survival Hypothesis: Combined PD-1 blockade with pembrolizumab + epacadostat in HNSCC patients will lead to improved 1-year survival in patients who a) progress on prior anti-PD-1/PD/L1 therapy on, and/or b) compared to patients who progress on 2nd line chemotherapy.
2. Safety Hypothesis: Combined treatment with pembrolizumab and epacadostat will be safe and tolerable in HNSCC patients.

Exploratory/Translational Objectives

1. Interferon-gamma Gene Expression Profile (GEP) (Seiwert ASCO 2015, Ribas ASCO 2015) and evaluation of RR, PFS, and OS in GEP positive and GEP negative patients.
2. Determine the micro-environment that underlies resistance/suboptimal treatment

   1. underlying degree of tumor inflammation
   2. Baseline PD-L1 expression

   d) Determine underlying Interferon Gamma signature
3. Assess underlying mutational burden (Snyder 2014)) Preclinical hypothesis: IDO1 inhibition will alter the micro-environment to a be "more T-cell inflamed" and make tumors amenable to benefit from anti-PD-1 treatment (when given concurrently with IDO1 inhibition). Hence we will evaluate tumors, with prior response exhibiting acquired resistance as well as tumors with minor/suboptimal benefit from prior PD-1/PD-L1 therapy for evidence (at baseline) of suboptimal immune microenvironmental conditions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have histologically confirmed squamous cell carcinoma of the head and neck (unresectable and not amenable to curative intent therapy)
* 2. Meet criteria for either the Acquired Resistance OR the Suboptimal Benefit Cohort

  a. Acquired Resistance is defined as (i and ii must both be met): i. Prior benefit from anti-PD-1/PD-L1 therapy defined as a) prior response, and/or b) ≥5 months of stable disease (SD). Intervening therapies are allowed.

ii. Progressive Disease (PD) on recent scans b. Suboptimal Benefit is defined as (i and ii must both be met): i. Prolonged stable disease ≥5 months OR Suboptimal response (>10% & <50% shrinkage per RECIST at any evaluation timepoint) ii. Ongoing stable disease on recent scans iii. Last treatment with an anti-PD-1/PD-L1 agent within 6 weeks prior to starting protocol treatment

* 3. Archival tissue for PD-L1 staining (alternatively a new biopsy (core) at baseline can be used). A minimum of 10 slides is required (unless approval from the PI is obtained)
* 4. Measurable disease per RECIST 1.1.
* 5. Known HPV status
* 6. ECOG performance status 0 or 1
* 7. Be willing and able to provide written informed consent/assent for the trial.
* 8. Be greater than or equal to 18 years of age on day of signing informed consent.
* 9. Demonstrate reasonable organ function as defined below, all screening labs should be performed within 10 days of treatment initiation.

System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculateda creatinine clearance ≤1.5 X upper limit of normal (ULN) OR (GFR can also be used in place of creatinine or CrCl) ≥40 mL/min for subject with creatinine levels > 2.0 X institutional ULN Hepatic Serum total bilirubin ≤ 1.2 X ULN OR in case of Gilbert's disease an elevated total Bilirubin is allowed if direct Bilirubin is ≤40% of total AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN

Coagulation International Normalized Ratio (INR) or Prothrombin Time ≤1.5 X ULN unless subject is receiving (PT) anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

*Creatinine clearance should be calculated per institutional standard.

* 10. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* 11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* 12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* 1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks of the first dose of treatment.
* 2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* 3. Has a known history of active TB (Bacillus Tuberculosis)
* 4. Has hypersensitivity to pembrolizumab, epacadostat or any of its excipients.
* 5. Has had a prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1, or targeted small molecule therapy within 2 weeks prior to study Day 1, or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* 6. Has not recovered from prior surgery, chemotherapy or radiation therapy from adverse events due to a previous treatment/ administered agent (i.e., ≤ Grade 1 or return to baseline prior to treatment).

Note: Subjects with ≤ Grade 2 neuropathy, any grade hearing loss or tinnitus, or typical side effects from radiotherapy are an exception to this criterion and may qualify for the study.

Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

* 7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence live expectancy in the subsequent 3 years without active treatment (e.g. low grade prostate cancer in absence of therapy).
* 8. Has known active (=growing) central nervous system (CNS) metastases and/or carcinomatous meningitis. Radiation or resected brain metastasis are acceptable if clinically stable.
* 9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* 10. Has known history of, or any evidence of active, non-infectious pneumonitis.
* 11. Warfarin use, even if low dose warfarin is not acceptable. However, other anti-coargulants (e.g. aspirin, enoxaparin and heparin derivatives, thrombin inhibitors, etc) are acceptable.
* 12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* 13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* 14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* 15. Has received prior therapy with an IDO inhibiting agent.
* 16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* 17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* 18. Has received a live vaccine within 30 days of planned start of study therapy.
* 19. Subjects receiving MAO-inhibitors (MAOI) or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening.
* 20. Any history of Serotonin Syndrome after receiving serotonergic drugs.
* 21. History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful. Screening QTc interval > 470 milliseconds is excluded. In the event that a single QTc is > 470 milliseconds, the subject may enroll if the average QTc for the 3 ECGs is < 470 milliseconds. For subjects with an intraventricular conduction delay (QRS interval > 120 milliseconds), the JTc interval may be used in place of the QTc with sponsor approval. The JTc must be < 340 milliseconds if JTc is used in place of the QTc. Subjects with left bundle branch block are excluded.

Note: QTc prolongation due to pacemaker may enroll if the JTc is normal.

* 22. Use of any UGT1A9 inhibitor from screening through follow-up period, including the following: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid.
* 23. History of organ transplant that requires use of immunosuppressives.
* 24. Any condition that would jeopardize the safety of the subject or compliance with the Protocol.
* 25. Clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, and arrhythmia requiring therapy Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed within 30 days prior to initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Patient response rate | From the start of treatment to the time of response until disease progression, death, or end of trial, whichever comes first, not to exceed 5 years.
  The number of patients with responses per RECIST 1.1 will be compared to the total number of patients in each cohort (which is anticipated to enroll 15).

SECONDARY OUTCOMES:
Overall survival rate | From the time of enrollment until death, withdrawal of consent, or the end of the study, whichever occurs first OR at most 2 years out from the last patient receiving treatment.
One year progression free rate | From the time of enrollment until the first documented disease progression, death, withdrawal of consent, or the end of the study, whichever occurs first OR at most 2 years out from the last patient receiving treatment.
Number of patients with adverse events | From the start of treatment until the end of study, not to exceed 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States